CLINICAL TRIAL: NCT05193149
Title: Reducing Exercise Intolerance Through Inspiratory Muscle Training in Obese Breast Cancer
Brief Title: Inspiratory Muscle Training in Obese Breast Cancer Survivors
Acronym: IMOCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Dharini Bhammar, Assistant Professor, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OSU-22220
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cancer Survivors; Obesity; Breast Cancer
MeSH Terms: conditions — Obesity; Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Staff completing outcomes testing and study participants will be blinded to treatment assignment (IMT/SHAM). The IMT/SHAM devices are the same with ability to alter resistance; however, upon use at the lower intensity, the participant may be able to tell whether the device has resistance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4 wk IMT + 12 wk exercise (Experimental): 4 weeks of IMT, 3/week, 3 sets of 15 repetitions, intensity up to 70% of MIP using a pressure threshold device PLUS 12 weeks of aerobic exercise training including cycling, walking, elliptical, starting in week 5, 3/week, up to 50min per session, moderate intensity
  Interventions: Behavioral: Inspiratory muscle training; Behavioral: Exercise training
- 4 wk SHAM + 12 wk exercise (Sham Comparator): 4 weeks of SHAM training, 3/week, 3 sets of 15 repetitions, intensity up of 10% of MIP using a pressure threshold device PLUS 12 weeks of aerobic exercise training including cycling, walking, elliptical, starting in week 5, 3/week, up to 50min per session, moderate intensity
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Inspiratory muscle training — Training of respiratory muscles
  Arms: 4 wk IMT + 12 wk exercise
Behavioral: Exercise training — Supervised aerobic exercise intervention

SUMMARY:
The investigators propose a randomized controlled trial to determine the effectiveness of inspiratory muscle training in improving exercise tolerance among stage 0-III obese breast cancer survivors.

DETAILED DESCRIPTION:
Randomized controlled trial (RCT) where obese participants (N=133) are randomized to 2 arms: [i] IMT 4 wks + Exercise 12 wks, [ii] SHAM 4 wks + Exercise 12 wks).

ELIGIBILITY:
Inclusion Criteria:

* completed active treatment for a Stage 0-III breast cancer diagnosis within 6 months to 5 years of enrollment.
* obese as defined by a body mass index (BMI) of 30 to 50 kg/m2
* patients who are on adjuvant endocrine therapy will be allowed to participate.
* sedentary (participating in less than 90 min of moderate intensity activity per week) and have at least one limitation in activity on the 10-question RAND-36 Physical Function Subscale to ensure some exercise intolerance

Exclusion Criteria:

* functional limitations that make independent exercise unsafe
* metastatic breast cancer
* ongoing or active infection with recent antibiotics or steroids
* Bilateral Axillary lymph node dissection (ALND) of >5 lymph nodes on each side, which could increase risk of lymphadenopathy with repeated blood pressure measurements during exercise or if patient has been advised by their clinician to avoid repeated BP measures on both arms. Bilateral Sentinel Lymph Node Biopsy (SLNB) will be allowed.
* heart disease precluding exercise (congestive heart failure, unstable angina pectoris, cardiac arrhythmia)
* psychiatric illness/social situations that would limit compliance with study requirements
* orthopedic or neuromuscular disorders or arthritis that preclude participation in exercise
* unwilling or unable to follow protocol requirements
* pregnant or nursing
* any condition which in the investigator's opinion deems the subject an unsuitable candidate to participate in this study
* presence of provokable ECG changes suggestive of heart disease, or dangerous arrhythmias or exercise induced hypertension, etc. during the cardiopulmonary exercise test
* non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in exercise tolerance | Baseline to 4 weeks
  Continuous variable assessed as time to exhaustion during a CWRET at 80% of peak work rate. Units: minutes.
Change in exercise tolerance | Baseline to 16 weeks
  Continuous variable assessed as time to exhaustion during a CWRET at 80% of peak work rate. Units: minutes.

SECONDARY OUTCOMES:
Change in inspiratory muscle strength | Baseline to 4 weeks
  Continuous variable, Maximal inspiratory pressure. Units: cm H20
Change in inspiratory muscle strength | Baseline to 16 weeks
  Continuous variable, Maximal inspiratory pressure. Units: cm H20
Change in inspiratory muscle endurance | Baseline to 4 weeks
  Continuous variable, Maximal voluntary ventilation in 12 seconds. Units: L/min
Change in inspiratory muscle endurance | Baseline to 16 weeks
  Continuous variable, Maximal voluntary ventilation in 12 seconds. Units: L/min
Change in exercise capacity | Baseline to 4 weeks
  Continuous variable, peak oxygen uptake. Units: L/min
Change in exercise capacity | Baseline to 16 weeks
  Continuous variable, peak oxygen uptake. Units: L/min
Change in dyspnea | Baseline to 4 weeks
  Continuous variable, mMRC dyspnea scale score. Units: score 0 to 4
Change in dyspnea | Baseline to 16 weeks
  Continuous variable, mMRC dyspnea scale score. Units: score 0 to 4
Change in fatigue | Baseline to 4 weeks
  Continuous variable, FACIT:F version 4 total score. Units: score 0 to 52
Change in fatigue | Baseline to 16 weeks
  Continuous variable, FACIT:F version 4 total score. Units: score 0 to 52

CONTACTS AND LOCATIONS:
Overall Officials: Dharini M Bhammar, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make deidentified data freely available if requested. The privacy and rights of the participants will be protected.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after data collection is complete for up to 3 years.
Access Criteria: Deidentified data will be made available on request following approved data use agreements between institutions.

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu